CLINICAL TRIAL: NCT06702072
Title: Change in Task-related Oxygen Uptake After Bronchoscopic Lung Volume Reduction With Endobronchial Valves
Brief Title: Change in Task-related Oxygen Uptake After EBV Treatment
Acronym: CROCODILE
Status: Not yet recruiting | Type: Observational
Sponsor: Dirk-Jan Slebos (Other)
Responsible Party: Sponsor-Investigator, Dirk-Jan Slebos, MD PhD, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Other Study IDs: CROCODILE
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: COPD
Keywords: COPD; Emphysema; lung volume reduction; endobronchial valves; bronchoscopy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endobronchial valve treatment: Patients who are undergo a bronchoscopic treatment using endobronchial valves.
  Interventions: Device: Endobronchial valve treatment

INTERVENTIONS:
Device: Endobronchial valve treatment — Endobronchial valve treatment

SUMMARY:
Rationale: Bronchoscopic lung volume reduction using endobronchial valves (EBV) has emerged as a viable treatment option for eligible patients with severe emphysema. In all studies conducted so far, exercise capacity has only been measured using the 6-minute walk distance test (6MWT). It is known that patients with COPD frequently experience problems during ADL, which can lead to avoidance of or care dependency for performing certain tasks and have a significant social impact on their lives.

Patients report that it is easier to perform ADLs after EBV treatment. Previously it was found that it was easier for patient to perform these activities after the EBV treatment. However, the physiological load during these ADLs has never been investigated before.

Potentially, EBV treatment could improve the metabolic load and consequently symptom perception, thus enhancing the execution of ADLs, which is an important patient-centred outcome. However, this has not been investigated so far.

Objective: To investigate the change in exercise physiology during daily activities after EBV treatment.

Study design: Observational study in which the study population will be asked to perform some additional test during regular visits for the bronchoscopic lung volume reduction treatment with valves.

Study population: Patients with emphysema who are scheduled for a bronchoscopic lung volume reduction treatment using endobronchial valves.

Intervention: Not applicable Main study parameters: The change in task-related oxygen uptake measured with a mobile oxygen device during activities of daily life 6 months after EBV treatment.

DETAILED DESCRIPTION:
Rationale: Bronchoscopic lung volume reduction using endobronchial valves (EBV) has emerged as a viable treatment option for eligible patients with severe emphysema. In all studies conducted so far, exercise capacity has only been measured using the 6-minute walk distance test (6MWT). The 6MWT is conducted under laboratory conditions, which weakly correspond to activities of daily living (ADL). It is known that patients with COPD frequently experience problems during ADL, which can lead to avoidance of or care dependency for performing certain tasks and have a significant social impact on their lives.

Patients report that it is easier to perform ADLs after EBV treatment. Previously, it was found that it was easier for patient to perform these activities after the EBV treatment. However, the physiological load during these ADLs was not investigated before. This could be measured with a mobile oxygen device which can measure oxygen uptake (VO2) and carbon dioxide production (VCO2) under more functional conditions and thus measure the metabolic load of these activities.

Potentially, EBV treatment could improve the metabolic load and consequently symptom perception, thus enhancing the execution of ADLs, which is an important patient-centred outcome. However, this has not been investigated so far.

Objective: To investigate the change in exercise physiology during daily activities after EBV treatment.

Study design: Observational study in which the study population will be asked to perform some additional test during regular visits for the bronchoscopic lung volume reduction treatment with valves.

Study population: Patients with emphysema who are scheduled for a bronchoscopic lung volume reduction treatment using endobronchial valves.

Intervention: Not applicable Main study parameters: The change in task-related oxygen uptake measured with a mobile oxygen device during activities of daily life 6 months after EBV treatment.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This study has no specific benefits for the participating patients and the study also has no major risks.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is scheduled for a bronchoscopic lung volume treatment using Pulmonx Zephyr Endobronchial Valves;
2. Patient read, understood and signed the Informed Consent Form.

Exclusion Criteria:

1) Patients who cannot perform ADL activities without the use of Long Term Oxygen Therapy (LTOT).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population exists of patients with severe emphysema who undergo a bronchoscopic lung volume reduction treatment with one-way endobronchial valves.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Task-related oxygen uptake | 6 months follow up
  The change between baseline and 6 months of follow up after EBV treatment in task-related oxygen uptake (VO2) during a set-up daily life activity trail.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Depends on the request